CLINICAL TRIAL: NCT01534845
Title: A Randomized Phase 2 Study to Evaluate the Efficacy Between Only Radiotherapy Versus CCRT With Temozolomide in Newly Diagnosed Grade III Gliomas Without 1p/19q Codeletion
Brief Title: Efficacy Study of Radiotherapy Alone Versus CCRT With Temozolomide in Grade III Gliomas Without 1p/19q Codeletion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jong Hoon Kim (Other)
Responsible Party: Sponsor-Investigator, Jong Hoon Kim, Professor, Department of Neurological Surgery, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNOG-1101
Record Dates: First submitted 2012-02-06; First posted 2012-02-17 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Anaplastic Glioma of Brain; Loss of Chromosomes 1p/19q
MeSH Terms: interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- only Radiotherapy (No Intervention): fractionated focal irradiation in daily fractions of 2 Gy given 5 days per week for 6 weeks, for a total of 60 Gy
- CCRT with Temozolomide (Active Comparator): RT with daily temozolomide (75 mg/m2/day, 7 days/week) from the first to the last day of radiotherapy) and adjuvant TMZ chemotherapy (150-200 mg/m2 po qd for 5 days q 28 days for 6 cycles).
  Interventions: Drug: Temozolomide (Temodal)

INTERVENTIONS:
Drug: Temozolomide (Temodal) — RT with daily temozolomide (75 mg/m2/day, 7 days/week) from the first to the last day of radiotherapy) and adjuvant TMZ chemotherapy (150-200 mg/m2 po qd for 5 days q 28 days for 6 cycles)
  Other Names: Temodal
  Arms: CCRT with Temozolomide

SUMMARY:
1. The management of anaplastic gliomas of WHO grade 3 is currently largely based on surgery followed by radiotherapy, of which prognosis remains still dismal with the median survival of 2-5 years. To date, the benefit of chemo for WHO grade 3 gliomas is unclear of modest at best with conventional cytotoxic agents, and the role of temozolomide for these entities still is not elucidated.
2. Codeletion of chromosome 1p/19q is considered the most important marker of prognostic significance in WHO grade 3 gliomas.
3. To project a randomized phase 2 screening trial examining the efficacy of concurrent chemoradiotherapy with temozolomide followed by adjuvant temozolomide for WHO grade 3 gliomas without codeletion of chromosome 1p/19q.
4. The prognostic significance of methylation status of MGMT and IDH1 mutation as molecular markers will be also assessed in each arm as key secondary analysis.

DETAILED DESCRIPTION:
The role of chemotherapy for gliomas has been recently reappraised by the advent of temozolomide, especially for glioblastomas, and further investigation is now being directed to unveiling its optimal indications, dosing protocols, and the most relevant prognostic factors. Meanwhile, the management of anaplastic gliomas of WHO grade 3 (anaplastic astrocytomas, anaplastic oligodendrogliomas, and anaplastic oligoastrocytomas) is currently largely based on surgery followed by radiotherapy, of which prognosis remains still dismal with the median survival of 2-5 years. To date, the benefit of chemo for WHO grade 3 gliomas is unclear of modest at best with conventional cytotoxic agents, and the role of temozolomide for these entities still is not elucidated. Moreover, WHO grade 3 gliomas are now known to consist of heterogeneous groups of different histologic features, biological behaviors, and prognoses. Accordingly, relevant molecular markers are appreciated with the growing body of data that showing their implications on response to therapy and survival, including codeletion of chromosome 1p/19q, methylation status of methylguanine methyl transferase (MGMT), and isocitrate dehydrogenase (IDH) mutation.1,4-6,11 Among those, codeletion of chromosome 1p/19q is considered the most important marker of prognostic significance in WHO grade 3 gliomas.

One recent Korean prospective cohort study showed the potential survival benefit and safety of concurrent chemoradiotherapy with temozolomide followed by adjuvant temozolomide for WHO grade 3 gliomas. In this study, however, the role of molecular markers such as codeletion of chromosome 1p/19q and MGMT methylation could not be determined because of small number of patients available. These results prompted this Korean group to project a randomized phase 2 screening trial examining the efficacy of concurrent chemoradiotherapy with temozolomide followed by adjuvant temozolomide for WHO grade 3 gliomas without codeletion of chromosome 1p/19q. The basic concept of the present clinical trial is "a subgroup with expected worse prognosis according to the status of chromosome 1p/19q, i.e. one without codeletion of chromosome 1p/19q is to be managed more aggressively", to investigate the role of temozolomide. An aggressive therapy (surgery + concurrent chemoradiotherapy with temozolomide followed by adjuvant temozolomide) will be compared to the conventional arm (surgery + radiotherapy only) in terms of its efficacy and safety for WHO grade 3 gliomas without chromosome 1p/19q codeletion. The prognostic significance of methylation status of MGMT and IDH1 mutation as molecular markers will be also assessed in each arm as key secondary analysis. Until now, there have been no such trials examining the efficacy and safety of temozolomide for WHO grade 3 gliomas based on prospective molecular stratification.

ELIGIBILITY:
Inclusion criteria:

* Newly diagnosed histologically proven supratentorial anaplastic gliomas.The histological diagnosis must be obtained from a neurosurgical resection or biopsy of a tumor including an open biopsy or stereotactic biopsy.
* Absence of chromosome 1p/19q co-deletion
* Age 18 years
* Eastern Cooperative Oncology Group performance status of 0-1
* Stable or decreasing dose of steroids for 5 days prior to randomization
* Meets 1 of the following RPA classifications:class III-V
* Adequate hematologic, renal, and hepatic function
* Written informed consent

Exclusion criteria:

* Prior chemotherapy within last 5 years
* Prior radiotherapy of the head and neck area
* Receiving concurrent investigational agents or has received an investigational agent within 30 days prior to randomization
* Planned surgery for other diseases (e.g. dental extraction)
* History of malignancy. Subjects with curatively treated cervical carcinoma in situ or basal cell carcinoma of the skin, or subjects who have been free of other malignancies for 5 years are eligible for this study
* Pregnant or lactating women
* Subject who disagree to follow acceptable methods of contraception
* Concurrent illness including unstable heart disease despite appropriate treatment, history of myocardial infarction within 6 months, serious neurological or psychological disease, and uncontrolled infection
* Subject unable to undergo Gd-MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-03; Primary Completion 2015-02 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
2-year progression free survival(PFS) | Assessed and followed for the duration of hospital stay, an expected average of 3 months
  Final primary end-point: 2 year PFS. Progression free survival(PFS) is defined as the time from randomization to progressive disease or death, which ever occurs earlier.

SECONDARY OUTCOMES:
5-year overall survival (OS) | assessed at 10 wks, 22 wks, 34 wks, and followed up every 4 months until documentation of death.
  final secondary end-point : 5-year OS. Overall survival is defined as the time from randomization to death, which ever occurs earlier.
5-year progression-free survival (PFS) | assessed at 10 wks, 22 wks, 34 wks, and followed up every 4 months until documentation of disease progression or death.
  final end-point : 5-year PFS
Safety (adverse events) | up to 5 years
Methylation status of MGMT | baseline
  confirmed by MS-PCR.
IDH mutation | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hoon Kim, Professor, Principal Investigator — Asan Medical Center; Jae Young Kim, professor, Study Director — SNUH
Locations (1):
- Asan Medical Center, Seoul, South Korea